CLINICAL TRIAL: NCT05538728
Title: A Prospective Open-label Study to Evaluate Safety and Effectiveness of Two Different Reconstitution Volumes of Poly-l-lactic Acid (PLLA) for Correction of Wrinkles in the décolletage Area
Brief Title: An Open-label Study of Poly-l-lactic Acid for Correction of Wrinkles in the décolletage Area
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 43USSA2112
Record Dates: First submitted 2022-09-08; First posted 2022-09-14 (Actual); Results first posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Wrinkles in Decolletage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- 8ml (Active Comparator): Device: Sculptra current label dilution for treatment of wrinkles in the decolletage area
  Interventions: Device: poly-l-lactic acid (Sculptra)
- 17ml (Active Comparator): Experimental: PLLA new dilution volume for treatment of wrinkles in the decolletage area
  Interventions: Device: poly-l-lactic acid (Sculptra)

INTERVENTIONS:
Device: poly-l-lactic acid (Sculptra) — Sculptra

SUMMARY:
This is a prospective open-label study to evaluate safety and effectiveness of two different reconstitution volumes of poly-l-lactic acid (PLLA) for correction of wrinkles in the décolletage area.

DETAILED DESCRIPTION:
A challenge for wrinkle correction of the decolletage/chest and other non-facial areas is that larger surface areas typically need to be treated than for facial indications, for which reason the Sponsor is investigating a larger reconstitution volume compared to the approved label. In this study, the total volume of 18mL, including 1mL of 2% lidocaine, is being explored and compared with results from the current labeled volume of 9mL, including lidocaine, to assess if the larger volume is well-tolerated for treatment for wrinkles in the decolletage area.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant, non-breastfeeding females over the age of 22
* subjects seeking treatment for the décolletage
* subjects with moderate (Grade 2) or severe (Grade 3) on the Galderma Décolletage Scale
* subjects willing to abstain from any other surgical or cosmetic procedures in the décolletage area for the duration of the study.

Exclusion Criteria:

* Known/previous allergy or hypersensitivity to Sculptra
* Previous tissue augmenting therapy, contouring or revitalization treatment in the décolletage prior to baseline
* Any plastic surgery or permanent surgical implant in the treatment area
* Previous treatment/procedure in the treatment area in the previous 6 months that would interfere with study injections or study assessments

Min Age: 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Galderma R&D
Locations (2):
- United States (2):
  - Galderma Study Site, Encino, California
  - Galderma Study Site, Solana Beach, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at the United States from 31 August 2022 to 08 August 2023.
Pre-assignment Details: A total of 30 participants were enrolled and treated in this study.
Groups:
- Sculptra 8ml: Participants received first treatment injection sub-dermally with Sculptra 8 milliliters (ml; current labeled total volume: reconstituted with 8 mL sterile water for injection [SWFI] + 1 mL lidocaine hydrochloride 2 percent [%]) at Day 1. After first treatment, if needed, an additional 3 treatment sessions were performed at 1 month (+ 2 weeks) interval. Treatment was continued till optimal correction, which was defined as at least one grade improvement on Galderma Decolletage Scale (GDS) and best correction that achieved as agreed upon by the Treating Investigator and the participant.
- Sculptra 17ml: Participants received first treatment injection sub-dermally with Sculptra 17ml (reconstituted with 17 mL SWFI + 1 mL lidocaine hydrochloride 2%) at Day 1. After first treatment, if needed, an additional 3 treatment sessions were performed at 1 month (+ 2 weeks) interval. Treatment was continued till optimal correction, which was defined as at least one grade improvement on GDS and best correction that achieved as agreed upon by the Treating Investigator and the participant.
Period: Overall Study
Arm/Group | Sculptra 8ml | Sculptra 17ml
Started | 16 | 14
Completed | 15 | 13
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population Included all participants who were randomized and analyzed according to the treatment they were randomized based on the randomization scheme.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sculptra 8ml | Sculptra 17ml | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (9.77) | 55.0 (8.88) | 54.0 (9.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 13 | 12 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 13 | 27
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders on the Galderma Décolletage Scale (GDS), as Assessed Live by the Treating Investigator, at Month 9
Description: Responder was defined as participants having at least one grade improvement from baseline. GDS was a validated 5-point scale used to assess the severity of lines and wrinkles in the décolletage area: Grade 0 (none to minimal), Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (very severe). Higher score meant very severe lines and wrinkles in the décolletage area.
Time Frame: At Month 9
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | Sculptra 8ml | Sculptra 17ml
Number analyzed (Participants) | 16 | 14
percentage of Participants | 93.8 [69.8 to 99.8] | 78.6 [49.2 to 95.3]

2. Secondary Outcome: Percentage of Responders on the Galderma Décolletage Scale, as Assessed Live by the Treating Investigator, at Month 6
Description: as for outcome 1
Time Frame: At Month 6
Population: ITT population Included all participants who were randomized and analyzed according to the treatment they were randomized based on the randomization scheme. Here, "overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | Sculptra 8ml | Sculptra 17ml
Number analyzed (Participants) | 15 | 12
percentage of Participants | 93.3 [68.1 to 99.8] | 100 [73.5 to 100.0]

3. Secondary Outcome: Percentage of Responders Who Achieved At Least "Improved" on the Global Aesthetic Improvement Scale (GAIS) as Assessed by Participant at Months 6 and 9
Description: Responder was defined as participants achieving 'very much improved', 'much improved' or "Improved" on GAIS compared to baseline. The 7-graded GAIS was used by the participant to live assess the severity of lines and wrinkles by responding to the question: "Please choose the response below that best describes the overall change in the appearance of your upper chest area since you received the study treatment " by using the respective categorical scale as follows: Very Much Improved, Much Improved, Improved, No Change, Worse, Much Worse, Very Much Worse. In this outcome measure, percentage of participants who achieved at least 'Improved' on the GAIS assessed by participant at Months 6 and 9 were reported.
Time Frame: At Month 6 and 9
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | Sculptra 8ml | Sculptra 17ml
Number analyzed (Participants) | 15 | 12
percentage of Participants
  At Month 6 | 100 [78.2 to 100.0] | 100 [73.5 to 100.0]
  At Month 9 | 100 [78.2 to 100.0] | 91.7 [61.5 to 99.8]

4. Secondary Outcome: Percentage of Responders With At Least "Improved" on the Global Aesthetic Improvement Scale (GAIS) as Assessed by Treating Investigator at Months 6 and 9
Description: Responder was defined as participants achieving 'very much improved', 'much improved' or "Improved" on GAIS compared to baseline. The 7-graded GAIS was used by the Treating Investigator to live assess the severity of lines and wrinkles by responding to the question: "Please choose the response below that best describes the overall change in the appearance of your upper chest area since you received the study treatment " by using the respective categorical scale as follows; Very Much Improved, Much Improved, Improved, No Change, Worse, Much Worse, Very Much Worse. In this outcome measure, percentage of participants who achieved at least 'Improved' on the GAIS assessed by treating investigator at Months 6 and 9 were reported.
Time Frame: At Months 6 and 9
Population: ITT population Included all participants who were randomized and analyzed according to the treatment they were randomized based on the randomization scheme. Here, 'number analyzed, n' signifies participants evaluable for specified time points.
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | Sculptra 8ml | Sculptra 17ml
Number analyzed (Participants) | 15 | 13
percentage of Participants
  At Month 6: number analyzed (Participants) | 15 | 12
  At Month 6 | 100 [78.2 to 100.0] | 100 [73.5 to 100.0]
  At Month 9 | 100 [78.2 to 100.0] | 100 [75.3 to 100.0]

ADVERSE EVENTS:
Time Frame: From Day 1 up to end of study (Up to 11 months)
Description: Safety population Included all participants who were treated with Sculptra.
Arm/Group | Sculptra 8ml | Sculptra 17ml
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 5/16 | 4/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sculptra 8ml (N=16) | Sculptra 17ml (N=14)
Injection site nodule (General disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Application site dermatitis (General disorders) | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
SARS-CoV-2 test positive (Investigations) | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/28/NCT05538728/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/28/NCT05538728/SAP_001.pdf